Date:12/01/2020

National Clinical Trials #: NCT03631745

Study Title: Delivering Church-based Interventions to Reduce Stigma and Mental Health Treatment Disparities Among Latinos



# **Informed Consent**

Your church, along with others is participating in a new project called *Proyecto AMÉN*. The project is about bringing the church together to learn about ways parishioners can support one another through the stresses and challenges of life. The program will involve educational presentations and church activities that raise awareness about mental health and resources that are intended to encourage, bring hope, and promote well-being among individuals and families within your parish. The project is funded by the National Institute of Minority Health and Health Disparities, part of the National Institutes of Health. RAND Corporation, a non-profit research organization, is running the project.

### **PROCEDURES**

To better understand the needs of parishes and the impact of the program, we will be asking parishioners to complete surveys. You will receive a \$20 gift card for completing a survey today. If you complete another survey in 6 months, you'll receive a \$30 gift card and if you complete another survey in 12 months you'll receive a \$40 gift card.

Each survey will take about 30 minutes to complete. The surveys will ask questions about how long you've attended this church and some basic demographics. They will also ask about your attitudes and beliefs toward mental health problems, your experiences with mental health problems and your use of alcohol. You may skip any question you do not wish to answer.

At each survey, you will be asked to complete a form with your contact information. This information will only be used to help us remind you of project activities and remind you to take the surveys. At the end of the project, your contact information will be destroyed.

### [Intervention]

Participating churches will invite congregants to attend educational presentations (Mental Health 101) held by the NAMI, as well as parish activities that will provide opportunities to learn about mental health: As a participant in this project, we ask that you attend at least 3 of these sessions. You may receive reminders from RAND to attend.

# [Waitlist Control]

In about a year, some participating churches including this one will invite congregants to attend educational presentations, such as Mental Health 101 held by the National Alliance on Mental Illness (NAMI), as well as parish activities that will provide opportunities to learn about mental health, how to help friends or family who may need support for a mental health problem, and ways your parish may be a refuge for those affected by mental health challenges. You do not need to attend these sessions to participate in this project.

### RISKS AND BENEFITS

It is possible you may experience some discomfort answering some of the survey questions. Again, you may skip any question you do not want to answer. If you attend the educational workshops, it is possible you may feel some discomfort as well. You are free to leave at any time.

### **CONFIDENTIALITY**

We will keep your responses confidential. Nobody, including church staff, will find out your answers to the survey. Your information is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the project cannot share any information that may identify you in any legal proceedings unless you say it is okay. This protection covers federal, state, or local civil, criminal, administrative, legislative, or other proceedings.

If you share during the project that you plan to harm yourself or others, the Certificate <u>does not</u> stop this from being reported to the proper authorities which is required by law.

If you have further questions, please ask them now. The Frequently Asked Questions document contains information on how to contact if you have future questions. For questions about your rights as a participant, you can contact RAND at 866-697-5620 and reference study # 2018-0189.

# ENROLLMENT AND CONSENT TO PARTICIPATE FORM

I have read (or someone has read to me) the information in the consent form, which explains the nature and purpose of this study. I have been given a chance to ask questions, and have all my questions answered. By signing below, I agree to participate in the project.

| Signature | Date |
|-----------------------------|------|
| Printed Name of Participant | |

Approved for use Dec 2020-Dec 2022 (online version consent)

# **Proyecto AMÉN Informed Consent**



Your church, along with others is participating in a new project called *Proyecto AMÉN*. The project is about bringing the church together to learn about ways parishioners can support one another through the stresses and challenges of life. The program will involve educational presentations and church activities that raise awareness about mental health and resources that are intended to encourage, bring hope, and promote well-being among individuals and families within your parish. This project is a collaboration between RAND Corporation, a non-profit research organization, and NAMI, the National Alliance on Mental Illness.

#### **PROCEDURES**

Will be asking parishioners to complete surveys:

- You will receive a \$20 Walmart gift card for completing the first survey as soon as you complete it. If you complete another survey in 6 months, you'll receive a \$30 gift card and if you complete another survey in 12 months, you'll receive a \$40 gift card.
- Each survey will take about 30 minutes to complete.
- The surveys will ask questions about how long you've attended this church and some basic demographics. They will also ask about your attitudes and beliefs toward mental health problems, your experiences with mental health problems and your use of alcohol. You may skip any question you do not wish to answer.
- At each survey, you will be asked to complete a form with your contact information—this information will only be used to help us remind you of project activities and remind you to take the surveys. At the end of the project, your contact information will be destroyed.

# [Intervention]

Participating churches will invite congregants to attend educational presentations (Mental Health 101) held by the NAMI, as well as parish activities that will provide opportunities to learn about mental health:

• As a participant in this project, we ask that you attend at least 3 of these sessions. You may receive reminders from RAND to attend.

### [Waitlist Control]

In about a year, some participating churches including this one will invite congregants to attend educational presentation (Mental Health 101) held by NAMI, as well as parish activities that will provide opportunities to learn about mental health. You do not need to attend these sessions to participate in this project.

### **RISKS AND BENEFITS**

- It is possible you may experience some discomfort answering some of the survey questions. **Again, you may skip any question you do not want to answer.**
- If you attend the educational workshops, it is possible you may feel some discomfort as well. You are free to leave at any time.

### CONFIDENTIALITY

- We will keep your responses confidential—nobody, including church staff, will find out your answers to the survey.
- Your information is covered by a Certificate of Confidentiality. This means that the project cannot share any information that may identify you in any legal proceedings unless you say it is okay.
- If you share during the project that you plan to harm yourself or others, the Certificate does not stop this from being reported to the proper authorities which is required by law.
- If you have further questions, please ask them now. The Frequently Asked Questions document contains information on how to contact if you have future questions.
- For questions about your rights as a participant, you can contact RAND at 866-697-5620 and reference study # 2018-0189.

### PARTICIPATION AND WITHDRAWAL

- You do not have to answer any survey question you do not wish to answer.
- If you take part in the project now, you are still free to refuse to take part in the follow-up surveys.
- You do not have to attend any sessions you do not wish to attend.
- Your participation in this project is completely voluntary.